CLINICAL TRIAL: NCT04204577
Title: Three-arm Open Parallel Control Phase II Trial for Evaluation of Thermal Ablation Combined With Apatinib and PD-1 Antibody SHR-1210 for Advanced Liver Cancer
Brief Title: The Safety and Efficacy of Thermal Ablation Combined With Apatinib and Carilimub for Advanced Liver Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Professor, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2019-128-02
Record Dates: First submitted 2019-08-28; First posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: BCLC Stage B Hepatocellular Carcinoma; BCLC Stage C Hepatocellular Carcinoma
MeSH Terms: interventions — apatinib; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thermal ablation (No Intervention): Taking standard thermal ablation treatment. Its specific number and time interval depend on the patient's own condition and disease.
- Thermal ablation combined with apatinib (Experimental): Taking standard thermal ablation treatment. Its specific number and time interval depend on the patient's own condition and disease.
  Oral apatinib mesylate tablets, 250 mg, orally once a day. Take about half an hour after a meal (the daily dose should be as much as possible), and take it with warm water. Apatinib was discontinued 7 days before each thermal ablation treatment, and after the thermal ablation treatment, the patient's aminotransferase returned to normal and continued to take apatinib.
  Interventions: Drug: Apatinib Mesylate
- Ablation combined with apatinib and PD-1 antibody SHR-1210 (Experimental): Taking standard thermal ablation treatment. Its specific number and time interval depend on the patient's own condition and disease.
  Oral apatinib mesylate tablets, 250 mg, orally once a day. Take it with warm water about half an hour after a meal (the daily dose should be as much as possible). Apatinib was discontinued 7 days before each thermal ablation treatment, and after the thermal ablation treatment, the patient's aminotransferase returned to normal and continued to take apatinib.
  SHR-1210, 200mg, intravenous infusion for 30 minutes (including the time of the tube,the overall infusion time is not shorter than 20 minutes, no longer than 60 minutes), once every 2 weeks; the first dose with the apatite Simultaneous administration of PD, PD-1 injection is not affected by thermal ablation.
  Interventions: Drug: Apatinib Mesylate

INTERVENTIONS:
Drug: Apatinib Mesylate — Evaluation of the efficacy and safety of simple local ablation, local ablation combined with apatinib, local ablation combined with apatinib and PD-1 antibody SHR-1210 for advanced liver cancer.
  Other Names: SHR-1210
  Arms: Ablation combined with apatinib and PD-1 antibody SHR-1210; Thermal ablation combined with apatinib

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of simple local ablation, local ablation combined with apatinib, local ablation combined with apatinib and PD-1 antibody SHR-1210 for the treatment of advanced liver cancer.

DETAILED DESCRIPTION:
Primary liver cancer is a common malignant tumor in the world. Its pathogenesis is concealed and clinically asymptomatic. It is mostly in the middle and late stages of the disease. It is often combined with different degrees of cirrhosis. The liver function reserve is poor.About 80% of patients are in the first place. The operation has been lost at the time of diagnosis.

Primary liver cancer is not sensitive to conventional treatments such as radiotherapy and chemotherapy because of its unique tissue type. For advanced liver cancer, ablation combined with other systemic treatments is expected to alleviate the patient's condition, prolong the patient's survival time, and benefit more patients. The long-term clinical efficacy of tumor thermal ablation has been reported more, the basic conclusion is consistent, hat is, the 5-year survival rate of early stage tumors such as liver cancer less than 3cm is not inferior to surgical resection, or even better. Liver cancer is rich in blood supply and tumor blood vessels are dense. The formation and maintenance of these blood vessels requires pro-angiogenic signals, of which VEGFR is a key component. Apatinib is a small molecule tyrosine kinase inhibitor that inhibits VEGFR at very low concentrations. SHR-1210 is a humanized anti-programmed cell death receptor 1 antibody.

This study was designed to evaluate the efficacy and safety of simple local ablation, local ablation combined with apatinib, local ablation combined with apatinib and PD-1 antibody SHR-1210 for the treatment of advanced liver cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-80 years old;
2. Patients with primary hepatocellular carcinoma who are strictly in accordance with the clinical diagnostic criteria for the diagnosis and treatment of primary liver cancer (2017 edition) or confirmed by histopathology or cytology;
3. Child-Pugh A or B;
4. BCLC B-C;
5. Eastern Cooperative Oncology Group(ECOG) body condition within a week before enrollment score 0-2;
6. Life expectancy of at least 3 months;
7. Adequate main organ function:
8. Hemoglobin ≥90g/L. Absolute neutrophil count (ANC) ≥1,500/mm3. Platelets ≥50,000/ul. Albumin ≥29g/L. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) <3 the upper limit of normal (ULN). Total bilirubin (TBIL) ≤1.5 ULN. Creatinine ≤1.5 ULN.
9. Women of childbearing age (generally 15-49 years of age) are required to have a negative pregnancy test (serum or urine) within 14 days prior to enrollment, and will voluntarily use the appropriate method of contraception during the observation period and within 8 weeks after the last administration of the study drug; For men, appropriate methods of contraception should be used during the observation period and within 8 weeks after the last administration of the study drug.
10. Be willing and able to provide written informed consent for the study.

Exclusion Criteria:

1. History of liver transplantation.
2. Other anti-angiogenic drugs and (or PD-1) antibody drugs were used within 3 months prior to enrollment.
3. History of immunosuppressive drugs used for 14 days prior to the first use of SHR-1210, excluding nasal and inhaled corticosteroids or physiological doses of systemic steroid hormones(no more than 10 mg/day of turpentine or equivalent) Pharmacological doses of other corticosteroids) .
4. Subjects are allergic to Apatinib Mesylate Tablets, SHR-1210, pharmaceutical excipients, or other monoclonal antibodies.
5. Attenuated Live Vaccine in four weeks before study or during study.
6. Uncontrolled or symptomatic active central nervous system (CNS) metastases are known to present with clinical signs, cerebral edema, spinal cord compression, cancerous meningitis, pia mater disease, and/or progressive growth. Patients with a history of central nervous system metastasis or spinal cord compression who have been treated and who have been clinically stable after 4 weeks of discontinuation of anticonvulsants and steroids prior to the study's first dose may be enrolled in the study.
7. Peripheral neuropathy grade >1.
8. There are any active autoimmune diseases or a history of autoimmune diseases (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, Hyperthyroidism, decreased thyroid function; subjects with vitiligo or complete remission in childhood asthma, can be included without adult intervention after adult; asthma requiring medical intervention for bronchodilators cannot be included).
9. History of human immunodeficiency virus (HIV) infection or known to have acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV-DNA≥1000 IU/ml), hepatitis C (positive hepatitis C antibody, and higher HCV-RNA than the lower limit of detection of the analytical method) or in combination with hepatitis B and hepatitis C, patients requiring antiviral therapy during the study;
10. Cardiovascular disease with 6 months before enrollment: Myocardial infarction, severe/unstable angina, NYHA class 2 or higher cardiac dysfunction, poorly controlled arrhythmias (including QTcF interval men >450 ms, women >470 ms, QTcF interval calculated by Fridericia formula), symptomatic hyperemia Sexual heart failure, cerebrovascular accident (including transient ischemic attack or symptomatic pulmonary embolism)
11. High blood pressure, and can not be well controlled by antihypertensive drugs (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90 mmHg)
12. Abnormal coagulation (INR >1.5×ULN or activated partial thromboplastin time (APTT) >1.5×ULN), with bleeding tendency or receiving thrombolysis or anticoagulant therapy.
13. Hereditary or acquired bleeding and thrombosis trends, such as hemophilia, coagulopathy, thrombocytopenia, hypersplenism, etc.
14. Obvious hemoptysis in the first 2 months before the study or daily hemoptysis exceed 2.5ml.
15. Significant clinically bleeding symptoms or clear bleeding tendency within 3 months prior to the study, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood (++) and above, or vasculitis.
16. Artery/ venous thrombosis, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism,etc.
17. Long-term anticoagulant therapy with warfarin or heparin or antiplatelet therapy (aspirin ≥300 mg/day or clopidogrel ≥75 mg/day).
18. Severe infection within 4 weeks prior to first drug administration (eg, intravenous infusion of antibiotics, antifungal or antiviral drugs), or unexplained fever >38.5℃ during screening period/first drug administration.
19. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
20. Participated in any other drug clinical study within 4 weeks prior to first drug administration , or no more than 5 half-lives from the last study.
21. History of psychotropic substance abuse or drug abuse.
22. Serious physical or mental illness, laboratory abnormalities, increasing risk of participating in the study, interfere with the results of the study, and patients considered by the investigator to be unfit for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival(PFS) | Up to two years
  The period between the onset of treatment from the onset of treatment, the observation of disease progression, or the death of any cause.

SECONDARY OUTCOMES:
Objective response rate (ORR) according to RECIST 1.1 | Up to approximately two years
  The proportion of patients with tumor size reduction of a predefined amount and for a minimum time period.
Disease control rate(DCR) | Up to approximately two years
  The proportion of patients who had a best response rating of complete response， partial response, or stable disease.
Overall survival(OS) | Up to approximately two years
  Overall survival is defined as time from the start of treatment until death due to any reason.
Overall survival rate of 6 months and 12 months | 6 months and 12 months
  Overall survival rate of 6 months and 12 months.
Safety: incidence and grade of adverse events (AEs) and Serious adverse events (SAEs) assessed by NCI-CTCAE v4.03 | Up to approximately two years
  The incidence and grade of adverse events (AEs) and Serious adverse events (SAEs) assessed by NCI-CTCAE v4.03
Quality of life score(QOL) | Up to approximately two years
  Quality of life score(QOL)0-100

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yu, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No